CLINICAL TRIAL: NCT00001082
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Adefovir Dipivoxil (Bis-POM PMEA) in Prolonging Survival of HIV-Infected Individuals With a CD4+ Cell Count of <= 100/mm3 or With a CD4+ Cell Count Both > 100 and <= 200/mm3 and a Nadir CD4+ Cell Count of <= 50/mm3
Brief Title: The Safety and Effectiveness of Adefovir Dipivoxil in the Treatment of HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPCRA 039; 11589 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: Cytomegalovirus Infections; Antiviral Agents; CD4 Lymphocyte Count; Prodrugs; Survival; Adenine
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections | interventions — Carnitine; adefovir dipivoxil

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): Participants will receive adefovir dipivoxil and L-carnitine
  Interventions: Drug: Levocarnitine; Drug: Adefovir dipivoxil
- 2 (Experimental): Participants will receive adefovir dipivoxil placebo and L-carnitine.
  Interventions: Drug: Levocarnitine; Drug: Adefovir dipivoxil placebo

INTERVENTIONS:
Drug: Levocarnitine — 500 mg tablet taken orally daily
  Other Names: L-carnitine
Drug: Adefovir dipivoxil — 120 mg tablet taken orally daily
  Arms: 1
Drug: Adefovir dipivoxil placebo — Oral placebo tablet taken daily
  Arms: 2

SUMMARY:
To evaluate the safety and efficacy of adefovir dipivoxil in prolonging survival of patients with advanced HIV disease. In CMV prophylaxis substudy: To evaluate the efficacy of adefovir dipivoxil in preventing the development of CMV end-organ disease in patients with advanced HIV coinfected with CMV.

The optimal treatment for HIV infection and the prevention of CMV disease has not been identified. Currently available antiretroviral therapies are hampered by both significant toxicities and the development of resistance. In addition, agents for preventing CMV disease, such as oral ganciclovir, are complicated by poor bioavailability and decreased compliance secondary to toxicities. Moreover, discordant results have been reported regarding the effectiveness of oral ganciclovir for preventing CMV disease. There is a need for newer agents with anti-HIV and anti-herpesvirus activity that have good pharmacokinetic and safety profiles and that will be well tolerated by patients. Adefovir dipivoxil is an oral pro-drug of PMEA, a nucleoside analog with activity against a broad spectrum of retroviruses and herpesviruses, including important human pathogens, such as HIV-1, HIV-2 and CMV. Due to its anti-HIV and anti-herpesvirus activity, adefovir dipivoxil may be able to decrease the incidence of opportunistic herpesvirus infections and prolong survival in patients with advanced HIV infection.

DETAILED DESCRIPTION:
The optimal treatment for HIV infection and the prevention of CMV disease has not been identified. Currently available antiretroviral therapies are hampered by both significant toxicities and the development of resistance. In addition, agents for preventing CMV disease, such as oral ganciclovir, are complicated by poor bioavailability and decreased compliance secondary to toxicities. Moreover, discordant results have been reported regarding the effectiveness of oral ganciclovir for preventing CMV disease. There is a need for newer agents with anti-HIV and anti-herpesvirus activity that have good pharmacokinetic and safety profiles and that will be well tolerated by patients. Adefovir dipivoxil is an oral pro-drug of PMEA, a nucleoside analog with activity against a broad spectrum of retroviruses and herpesviruses, including important human pathogens, such as HIV-1, HIV-2 and CMV. Due to its anti-HIV and anti-herpesvirus activity, adefovir dipivoxil may be able to decrease the incidence of opportunistic herpesvirus infections and prolong survival in patients with advanced HIV infection.

All patients will be enrolled within the first 18 months of the study. They will be randomized to 1 of 2 groups. Group 1 will be comprised of 1080 patients and will receive adefovir dipivoxil plus L-carnitine and group 2 will be comprised of 1080 patients and will receive a placebo plus L-carnitine. At least the first 400 patients enrolled (200 in each group) will comprise the safety-HIV virology cohort. These patients will have more frequent follow up visits, additional laboratory evaluations, and more intensive safety data information during the first 6 months. NOTE: At least 850 patients who are infected with CMV are followed for the development of CMV end-organ disease in a CMV prophylaxis substudy.

AS PER AMENDMENT 8/7/97: All patients are enrolled in the primary study and randomized to the treatment or placebo regimen. Within the primary study, patients meeting specified criteria may be enrolled in one or more of the following cohorts:

1. Safety-HIV virology cohort (at least the first 400 patients enrolled in the study regardless of CMV status).
2. CMV bDNA cohort (those patients in the safety-HIV virology cohort who are CMV-positive).
3. CMV-virology cohort (the first 400 patients in the CMV bDNA cohort enrolled at sites able to obtain CMV urine cultures).

All patients who are CMV-positive are enrolled in the CMV prophylaxis substudy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chronically administered concomitant therapies for HIV and opportunistic diseases, including chemotherapy for cutaneous Kaposi's sarcoma, must be on these therapies for at least 30 days prior to study entry.
* Short courses of oral antibiotics or other therapies given for a limited period of 3 weeks.
* Episodic use of IV acyclovir or oral acyclovir > 1g/day for treatment of acute illness is permitted at the clinician's discretion.

Patients must have:

* A working diagnosis of HIV infection based on the patient's medical history, behavioral history, clinical signs and symptoms, or results of other laboratory tests.
* CD4+ cell count <= 100 cells/mm3 within 60 days prior to randomization (OR, AS PER AMENDMENT 8/7/97, a CD4+ cell count that is both > 100 and <= 200 cells/mm3 within 60 days prior to randomization and a documented nadir CD4+ cell count <= 50 cells/ mm3 at any time prior to randomization).
* Reasonably good health.
* Life expectancy of at least 6 months.
* Access to a refrigerator for the storage of adefovir dipivoxil.
* Signed informed consent from parent or legal guardian for patients less than 18 years of age.

AS PER AMENDMENT 8/7/97:

* CMV serology (IgG) positive (CMV bDNA cohort and CMV-virology cohort).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Evidence of active CMV disease at screening.
* Conditions that would require use of medications listed in Exclusion Concurrent Medications.

Concurrent Medication:

Excluded:

* Any investigational anti-CMV agent.
* Adenine arabinoside (vidarabine).
* Amantadine hydrochloride (Symmetrel).
* Cidofovir (Vistide).
* CMV hyperimmune globulin.
* Cytosine arabinoside (cytarabine).
* Famciclovir.
* Foscarnet (phosphonoformic acid).
* Ganciclovir (Cytovene).
* GW 1263W94 (Benzamidazole).
* Idoxuridine.
* Intravenous acyclovir.
* ISIS 2922 (Anti-sense).
* Lobucavir.
* MSL109.
* Oral acyclovir > 1 g/day.
* Valacyclovir.

Patients with the following prior conditions are excluded:

* History of CMV end-organ disease.

Prior Medication:

Excluded within 2 weeks of randomization:

* Any investigational anti-CMV agent.
* Adenine arabinoside (vidarabine).
* Amantadine hydrochloride (Symmetrel).
* Cidofovir (Vistide).
* CMV hyperimmune globulin.
* Cytosine arabinoside (cytarabine).
* Famciclovir.
* Ganciclovir (Cytovene).
* GW 1263W94 (Benzamidazole).
* Idoxuridine.
* Intravenous acyclovir.
* ISIS 2922 (Anti-sense).
* Lobucavir.
* MSL109.
* Oral acyclovir > 1 g/day.
* Valacyclovir.

Excluded within 60 days prior to study entry:

* Foscarnet.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 1996-12; Primary Completion 1999-01 (Actual); Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Morbidity | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Brosgart C, Study Chair; Fisher E, Study Chair
Locations (15):
- United States (15):
  - Community Consortium / UCSF, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Wayne State Univ - WSU/DMC / Univ Hlth Ctr, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research / New Mexico, Albuquerque, New Mexico
  - Harlem AIDS Treatment Grp / Harlem Hosp Ctr, New York, New York
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium / Div of Infect Diseases, Richmond, Virginia

REFERENCES:
- [Background] Fisher E, Brosgart C, Cohn D, Chaloner K, Pulling C, Alston B, Schmetter B, El-Sadr W. Placebo (PLC)-controlled, multicenter trial of adefovir dipivoxil (ADV) in patients (pt) with HIV disease. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:160 (abstract no 491)
- [Background] Brosgart C, Fisher E, Pulling C, Chaloner K, Cohn D, Elsadr W, Verheggen R, Schmetter B, Alston B. Prevalence of asymptomatic CMV retinitis (CMVR) in AIDS patients. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:152 (abstract no 453)
- [Background] Fisher E, Brosgart C, Cohn D, Chaloner K, Pulling C, Schmetter B, Alston B, El-Sadr W. Safety of adefovir dipivoxil (ADV) and incidence of proximal renal tubular disorder (PRTD) in a placebo (PLC)-controlled trial in patients (pt) with advanced HIV disease. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:195 (abstract no 678)
- [Background] Brosgart C, Pulling C, Chaloner K, Fisher E, Coakley D, Diggins M, Ivannidis J. Serum carnitine levels in AIDS patients with advanced HIV disease from the CPCRA 039 trial. Int Conf AIDS. 1998;12:1094 (abstract no 60508)